CLINICAL TRIAL: NCT00500188
Title: A Prospective, Randomized, Phase II Study of Preoperative Plus Postoperative Imatinib Mesylate (Gleevec, Formerly STI-571) in Patients With Primary, Recurrent, or Metastatic Resectable, Kit-Expressing, Gastrointestinal Stromal Tumor (GIST)
Brief Title: Preoperative and Postoperative Imatinib Mesylate Study in Patients With c-Kit Positive GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Jonathan Trent, MD, PhD/Assistant Professor, U.T.M.D. Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0023
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; GIST; Kit expression; Resectable; Imatinib Mesylate; Gleevec; STI-571; Imatinib; NSC-716051
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7 Days (Experimental): Imatinib Mesylate 300 mg orally twice daily starting 7 days before surgery.
  Interventions: Drug: Imatinib Mesylate (Gleevec)
- 5 Days (Experimental): Imatinib Mesylate 300 mg orally twice daily starting 5 days before surgery.
  Interventions: Drug: Imatinib Mesylate (Gleevec)
- 3 Days (Experimental): Imatinib Mesylate 300 mg orally twice daily starting 3 days before surgery.
  Interventions: Drug: Imatinib Mesylate (Gleevec)

INTERVENTIONS:
Drug: Imatinib Mesylate (Gleevec) — 300 mg orally twice daily
  Other Names: Gleevec; STI-571; Imatinib; NSC-716051

SUMMARY:
Primary objectives

1. To determine whether induction of apoptosis or inhibition of angiogenesis are involved in the antitumor activity of (Gleevec, Formerly STI-571) in patients with gastrointestinal stromal tumors (GIST) as assessed by Positron Emission Tomography (PET) scanning.
2. To determine whether dynamic computed tomography (CT), PET scan, molecular and histopathologic responses in GIST tumors from patients treated with Gleevec predict Disease-Free Survival (DFS) time.

Secondary objectives

1. To determine the disease free survival of patients with resectable or partially resectable gastrointestinal stromal tumors treated with Gleevec preoperatively and continued for 2 years after resection of disease.
2. To assess the safety and tolerability of Gleevec given to patients with GI stromal tumors 3, 5, or 7 days preoperatively and continued postoperatively.

DETAILED DESCRIPTION:
Imatinib mesylate is a drug that may help to kill gastrointestinal stromal tumor cells.

Around 3 weeks before your scheduled surgery, you will have a PET scan, a CT scan and two to three tablespoons of blood will be collected. These are imaging tests and are being done to check on the status of the disease. These tests will be repeated the day before your scheduled surgery. If your doctor feels it is necessary, you will have a chest x-ray and 2 to 3 tablespoons of blood will be collected for routine tests. Women who are able to have children must have a negative blood pregnancy test.

Before treatment, you will also have a biopsy procedure of the tumor performed. This biopsy is being done to study the effect of imatinib mesylate on the tumor cells. The tissue that is collected during the biopsy procedure will be compared to the tumor that is taken out at the time of surgery.

You will be randomly assigned (as in the toss of a coin) to one of three groups. One group will begin taking imatinib mesylate two times a day by mouth starting 7 days before surgery. The second group will start taking imatinib mesylate 5 days before surgery. Participants in the third group will begin taking imatinib mesylate 3 days before surgery. After your surgery, the removed tumor will be studied and compared to the tissue collected before surgery to see what effect (if any) imatinib mesylate had on the tumor. All patients will then continue imatinib mesylate for 2 years after surgery.

You will take imatinib mesylate two times a day for 2 years.

If you develop any side effects to the study drug, treatment may be temporarily stopped or the dose of the drug changed until the symptoms are gone. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

You will be seen by a physician regularly after surgery. Two to three tablespoons of blood will be collected once a month for routine tests, and a you will have a CT scan done every 3 months. These tests will help us determine if your cancer has come back.

THIS IS AN INVESTIGATIONAL STUDY. Imatinib mesylate is FDA approved and is commercially available. Up to 48 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Patients must have a histologically proven diagnosis of primary, locally advanced and/or metastatic GIST for which complete or partial resection is planned by a MDACC sarcoma surgeon.
3. Patients must have immunohistochemical documentation of kit expression in the tumor using the DAKO A4502 or other acceptable antibody.
4. Patients must have a least one lesion greater than 1 cm that can be accurately measured in one dimension by plain radiograph, CT or magnetic resonance imaging (MRI).
5. Patients must have normal organ and marrow function (White blood count-WBC greater than or equal to 3,000/ul, Absolute neutrophil count (ANC) greater than or equal to 1500/ul, platelets greater than or equal to 100,00/ul, total bilirubin less than or equal to 1.5 * Upper Limits of Normal (ULN), aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT) less than or equal to 2.5 * ULN, serum creatinine less than or equal to 1.5 * ULN).
6. Patients must have a serum glucose < 200 mg/dl prior to PET scan. Patients must be able to lie flat and still for the PET scan.
7. Patients may not have any uncontrolled medical or psychiatric conditions that would make the patient unable to tolerate therapy. Patients with uncontrolled medical conditions or psychiatric conditions may have informed consent granted by a legal guardian or surrogate decision maker.
8. Patients may not have any prior malignancy in the past 5 years other than non-melanoma skin cancer, cervical cancer in situ, or any other malignancy that is not currently clinically significant.
9. Zubrod performance status of 0 - 3.
10. May not have metastases outside of the peritoneal cavity.
11. If patients have any signs or symptoms of metastases, the appropriate workup should occur prior to enrollment (eg, CT of the head for a patient with central nervous system (CNS) symptoms).
12. Patients may not have had chemotherapy, radiotherapy, biological therapy or any investigational drugs 3 weeks prior to the study.
13. Women should have a negative pregnancy test within 7 days of study opening.
14. Patients must agree to use an effective contraceptive method.

Exclusion Criteria:

1. Prior treatment using Gleevec.
2. Patients with Class III or Class IV New York Heart Association congestive heart failure.
3. Pregnant or nursing women.
4. Patients taking therapeutic doses of Coumadin for anticoagulation. Coumadin may be taken but dose should be less than or equal to 1 mg po per day. Patients MAY take a low molecular weight heparin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) time | Baseline start of therapy to 2 years postoperative Gleevec or disease progression.
  Effect of drug imatinib mesylate on gastrointestinal stromal tumors (GIST) by disease-free survival (DFS) time, measured from the start of Gleevec therapy, among the three arms to disease progression or 2 years postoperative therapy, measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Trent, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org